CLINICAL TRIAL: NCT01481285
Title: Generation of Normal Ranges to Analyze Body Composition of Adults Based on Bioelectrical Impedance Analysis (BIA)
Status: Completed | Type: Observational
Sponsor: Seca GmbH & Co. Kg. (Industry)
Responsible Party: Sponsor
Other Study IDs: BCA-03 | BCA-04
Record Dates: First submitted 2011-07-21; First posted 2011-11-29 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: Bioelectrical Impedance Measurement; Adults

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- healthy adults: The study will cover 992 healthy adults. 496 men and 496 women in an age range of 18 to 65 years are planned to be recruited.

SUMMARY:
The aim of the study is to generate normal ranges for φ, BIVA and BCC. The calculation of FMI and FFMI is based on the results of two other clinical investigations: "Generation of prediction equation to analyze body composition of adults based on Bioelectrical Impedance Analysis (BIA)" (BCA-01) and "Application and adaption of device specific body composition formulas to various ethnic groups" (BCA-02). The aim of BCA-01 was to develop prediction equations for calculating FFM, TBW, ECW and SMM based on the gold standard reference methods ADP, DXA, MRI, D2O and NaBr on the one hand and measurement data of the BIA devices on the other hand. The equations are necessary to use the device as a Body Composition Analyzer with an acceptable accuracy level for clinical practice. The aim of the study BCA-02 was to apply and adapt device specific body composition formulas to various ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

The study will cover 992 healthy adults. 496 men and 496 women in an age range of 18 to 65 years are planned to be recruited. All subjects need to be suitable for blood donation according to "Hämotherapie-Richtlinie nach §§ 12a und 18 TFG", chapter 2.1.4 "Untersuchung zur Eignung als Spender und zur Feststellung der Spendertauglichkeit".

Exclusion Criteria:

* amputation of limbs
* electrical implant as cardiac pacemaker
* insulin pumps
* probands who cannot provide an ICF by themselves
* probands who might be dependent from the sponsor or the inv. site
* extensive tattoos at arms or legs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data of 992 healthy adults are planned to be collected.
Sampling Method: Probability Sample
Enrollment: 992 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Bioelectrical Impedance of 1, 1.5, 2, 3, 5, 7.5, 10, 15, 20, 30, 50, 75, 100, 150, 200, 300, 500, 750 and 1,000 kHz | about 15 minutes
  The measurement is planned to be done for all body segments: right arm, left arm, right leg, left leg, trunk, right body side and left body side. In total resistance and reactance at 19 frequencies for 7 body segments are planned to be measured.

SECONDARY OUTCOMES:
Verification of equivalence to a predicate device in accordance to Premarket Notification [510(k)] process of the FDA for product approval in the U. S. | about 15 minutes
  Predicate Device: BIOSPACE INBODY 720

CONTACTS AND LOCATIONS:
Overall Officials: Sven Peine, Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Institute for Transfusion Medicine, Hamburg, Hamburg, Germany

REFERENCES:
- [Derived] Enderle J, Reljic D, Jensen B, Peine S, Zopf Y, Bosy-Westphal A. Normal values for body composition in adults are better represented by continuous reference ranges dependent on age and BMI. Clin Nutr. 2023 May;42(5):644-652. doi: 10.1016/j.clnu.2023.03.006. Epub 2023 Mar 9. PMID 36933351